CLINICAL TRIAL: NCT02753829
Title: Home-based Cardiovascular Rehabilitation, Maintenance Phase, in Subjects With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ágata Sofia da Silva Vieira (Other)
Responsible Party: Sponsor-Investigator, Ágata Sofia da Silva Vieira, PHD Student, Universidade do Porto
Organization: Universidade do Porto (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASV-88
Record Dates: First submitted 2016-04-18; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Heart Disease; Acute Myocardial Infarction: Rehabilitation Phase
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental group 1 (Experimental): Cardiovascular rehabilitation program using Kinect of Xbox, in home care context,virtual format
  Interventions: Procedure: Cardiovascular rehabilitation program using Kinect of Xbox
- Experimental group 2 (Experimental): Cardiovascular rehabilitation program using paper manual, in home care context, conventional format
  Interventions: Procedure: Cardiovascular rehabilitation program using paper manual
- Control Group (Other): Educational component
  Interventions: Other: Educational component

INTERVENTIONS:
Procedure: Cardiovascular rehabilitation program using Kinect of Xbox — Participants perform a program of specific exercises. The exercise protocol was adapted to the home context and presented two progressive levels of intensity of exercise, having the second level being introduced after 3 months. The exercise protocol was performed at a moderate intensity, initiated, using data from the stress test, maximal heart rate, the Karvonnen formula, with 65% of the reserve heart rate, progressing for 70%.
  It was given the educational component about the control of cardiovascular risk factors and was encouraged to carry out the daily walks.
  Arms: Experimental group 1
Procedure: Cardiovascular rehabilitation program using paper manual — Participants perform a program of specific exercises. The exercise protocol was adapted to the home context and presented two progressive levels of intensity of exercise, having the second level being introduced after 3 months. The exercise protocol was performed at a moderate intensity, initiated, using data from the stress test, maximal heart rate, the Karvonnen formula, with 65% of the reserve heart rate, progressing for 70%.
  It was given the educational component about the control of cardiovascular risk factors and was encouraged to carry out the daily walks.
  Arms: Experimental group 2
Other: Educational component — It was only given the educational component about the control of cardiovascular risk factors and was encouraged to carry out the daily walks.
  Arms: Control Group

SUMMARY:
The sample of this randomized controlled trial was obtained in the Cardiovascular Prevention and Rehabilitation Unit, of the Hospital Centre of Porto, Santo Antonio General Hospital. The target population was individuals who have completed the training phase of cardiovascular rehabilitation program, volunteers and referenced by the responsible for the service.

This study has as main objective to analyze the influence of a specific exercise program, maintenance phase of cardiovascular rehabilitation , in home care context, for a period of 6 months, using a virtual format (computer and Kinect) or a conventional format (paper manual) in subjects with coronary artery disease. It was intended to analyze the immediate effect of exercise program on body composition and food consumption patterns, functional muscle strength of lower limb, level of physical activity: total volume of activity as well as the profile of this intensity, kyphotic index, balance, cognitive and executive function, as well as in the quality of life.

The aim is also to examine the effects, approximately 3 months after the end of the exercise program, in the lipid profile, the level of physical activity: total volume of activity as well as the profile of this intensity and cardiovascular fitness: maximum double product ; metabolic equivalents; and proof and recovery time.

The individuals were distributed at random, every 3 individuals, using the capabilities of Microsoft Excel 2010 RANDBETWEEN command, by three groups: the experimental group 1- a cardiovascular rehabilitation program, in home care context, using a computer and Kinect, virtual format, the experimental group 2- in cardiovascular rehabilitation program, in home care context, using a paper-based manual, conventional format, and control group-only subject to education for cardiovascular risk factors.

The program defined 3 training sessions per week. The rehabilitation program was oriented by the guidelines for exercise prescription.

Participants perform the a program of specific exercises independently and individually, with remote supervision, using communication (phone, email, etc.) and a routine scheduled individual meetings.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease diagnosed and stabilized
* both sexes
* aged between 40 and 75 years
* individuals were to have performed and completed the training phase of cardiovascular rehabilitation
* individuals should have a computer with at least Microsoft Windows 7

Exclusion Criteria:

* heart surgery
* individuals whose stress test did not end for maximum fatigue
* individuals in gestation period or wishing to become pregnant
* individuals classified as cardiovascular high-risk
* individuals with pacemakers or with severe neurological, musculoskeletal or respiratory diseases and metabolic unbalanced disease or reported dementia, cardiomyopathies, history of cardio respiratory arrest don't associated with acute myocardial infarction or cardiac procedures
* individuals with significant visual and auditory deficits not compensated
* individuals illiterate and / or without knowledge of Portuguese language
* Individuals who were in, or wanted to do gyms or other regular exercise programs during the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Cardiovascular fitness using the stress test | 9 months
Physical activity using the accelerometer | 9 months
Quality of life using Macnew (heart disease health-related quality of life questionnaire) | 6 months
Lipid Profile using laboratory tests | 9 months
Quality of life using EADS-21 (depression, anxiety and stress scale) | 6 months

SECONDARY OUTCOMES:
Balance using the One leg standing test | 6 months
Balance using Star Excursion Balance Test | 6 months
Kyphotic index using the flexicurve | 6 months
Cognitive function using the Trail Making Test | 6 months
Cognitive function using the Verbal Digit Span Test | 6 months
Cognitive function using the Stroop Test | 6 months
Weight using the balance of bioimpedance | 6 months
Total fat mass using the balance of bioimpedance | 6 months
Fat mass of the trunk using the balance of bioimpedance | 6 months
Lean body mass using the balance of bioimpedance | 6 months
Waist hip ratio using the tape measure | 6 months
Waist height ratio using the tape measure | 6 months
Food consumption patterns using the food frequency questionnaire | 6 months
Functional muscle strength of lower limb using the Sit-to-stand test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ágata S Vieira, Principal Investigator — Universidade do Porto

IPD SHARING:
Plan to Share IPD: No